CLINICAL TRIAL: NCT06859905
Title: The Effectiveness of Blood Flow Restriction Training on Upper Limb Motor Function, Strength, and Activity of Daily Living in Hemiparesis Post-stroke Patients
Brief Title: Blood Flow Restriction Training on Upper Limb Performance
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hail (Other)
Responsible Party: Principal Investigator, Ahmed Abdelmoniem Ibrahim, Associate Professor, University of Hail
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-2025-618
Record Dates: First submitted 2025-02-27; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Hemiparesis
Keywords: cerebro vascular accident, hemoplegia, blood restriction, performance, upper extremity
MeSH Terms: conditions — Paresis | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Intervention Model Description: The participants will be randomly divided into two groups: The study group low-load blood flow restriction training LIBFR(BFRT G), and control group (C G), all subjects in the control and BFRTG will receive the routine rehabilitation 3 times per week for 8 weeks
Who Masked: Outcomes Assessor
Masking Description: the participants will be allocated using the closed-envelop method with each envelop containing a card with a coded number. Particiants will be treated using these code numbers throughout the study. only the outcome assessor will not be allowed to have the interpritation of the coded numbers till the end of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- study group (Experimental): this group will receive blood flow restriction training (BFRT) plus regular exercises for the upper extremity for 8 weeks
  Interventions: Other: blood flow restriction training; Other: regular exercises
- control group (Active Comparator): this group will receive regular exercises for 8 weeks
  Interventions: Other: regular exercises

INTERVENTIONS:
Other: blood flow restriction training — Position of the patient The vascular occlusion pressure required for the full blockage of upper extremity blood flow will be measured at rest, with the individual relaxed in a sitting position(Sieljacks et al., 2018).
  Position of the of the cuff during BFRT
  Placing a 5 to 6 cm wide cuff on the more proximal part of the affected upper limb, it should be around the bulk of biceps muscle above the cubital fossa .
  BFRT Cuff Pressure The upper arm external pressure of the cuff (100-130 mmHg) will be selected concerning the subject's resting blood pressure as described previously by Yasuda et al. 2008 (Yasuda et al., 2008).
  BFRT exercises prescription
  1. Exercise frequency and duration
     -The study group (BFRT G) will be subjected to supervised exercises with low-load blood flow restriction training LIBFR (three days per week for 8 weeks),
  2. Exercise intensity -Low load blood flow restriction training LIBFR (20%-40% of 10 repetition maximum (10 RM) BFR training for the study group,
  Arms: study group
Other: regular exercises — the routine rehabilitation will be applied 3 times per week for 8 weeks, including the following training
  1. Appropriate neurodevelopmental techniques as needed by each patient
  2. Progressive resistance exercise for muscles in the affected upper extremity using sandbags, free weights, or elastic resistance bands according to each patient's abilities
  3. prolonged stretching using splints if needed
  4. Functional electrical stimulation (FES)

SUMMARY:
Background; Blood flow restriction training (BFRT) is a physical intervention that promotes many beneficial muscular activities and functions when low load/intensity is used in healthy and clinical populations.

Objectives: To determine the effect of BFRT on upper extremity motor function, strength, and Activity of daily living in chronic/acute stroke patients.

DETAILED DESCRIPTION:
A cerebrovascular accident (CVA) is often known as a stroke and can be described as a localized neurological deficiency caused by various cardiovascular abnormalities that disrupt brain function. Stroke is the primary cause of death worldwide, it also leads to a substantial number of disability among the population.

There is no doubt that stroke is one of the most common causes of adult-onset disabilities. 70-85% of the first strokes are associated with hemiplegia which is usually followed by hemiparesis. Only 60% of patients suffering from hemiparesis need physical rehabilitation and have attained functional independence in basic activities of daily living (ADLs) such as using the restroom and short-distance walking. Patients with sensorimotor and visual-field loss are much more dependent on care than those with pure motor impairments.

Stroke patients require post-stroke rehabilitation and physical therapy procedures to improve their recovery and quality of life. A multidisciplinary approach that addresses each patient's unique physical, occupational, and speech deficits can assist optimize their functional abilities and encourage independence.

Hemiplegic stroke rehabilitation involves structured, interdisciplinary, supportive services that start 48 hours after the stroke starts for stable patients. Although patients and families generally benefit from inpatient and outpatient rehabilitation, each treatment modality's efficacy falls short of standards set by evidence-based therapy (reference). Rehabilitation has always been around teaching patients how to compensate with their unaffected arm or limb. The major goals of physical, occupational, and speech therapists are to modify the surroundings and develop new skills in order to keep patients at home with the least amount of care assistance. The removal of architectural impediments to movement, problem-solving techniques, supporting social and psychological services, braces and other orthotics, and equipment like wheelchairs and walkers all continue to be crucial in assisting patients in doing daily life tasks (Dobkin, 2004).

The goal of physical therapy rehabilitation modalities post-stroke is to enhance activities of daily living, enhance range of motion, reduce pain, and improving muscle tone. Previous studies on BFRT have focused on healthy populations, limited number of observational trials have been performed on BFRT in patients with neurological problems, such as Parkinson's disease, multiple sclerosis, spinal cord injury, and stroke.

BFRT involves partially restricting arterial blood flow into muscles as well as occluding the venous outflow during exercise. It was first introduced into the literature by a Japanese doctor Yoshiaki Sato in Japan in 1987 who used tourniquet ischemia to induce muscle fatigue. This technique was originally called "kaatsu training," meaning "training with added pressure." Kaatsu training is now performed all over the world and is more commonly referred to as "BFRT" and is achieved using a pneumatic tourniquet system.

In addition to physical rehabilitation, BFRT is used for physical training and performance in healthy individuals. There has been extensive research into its value as a training tool, including elite- and amateur-level athletes, untrained young and older adults, and hypertensive individuals.

In addition to reducing arterial blood flow to working muscles, blood flow restriction obstructs venous return. When active muscles are exposed to BFR conditions, they are subjected to ischemia, which increases the metabolic stress on them. In addition to BFR, venous occlusion increases muscle cell swelling, activates intracellular anabolic pathways, and recruits fast-twitch fibers, which are thought to be involved in muscle adaptation.

There were different Factors affecting exercise adaptations with BFR including pressure of occlusion (partial or complete), type of occlusion (continuous or intermittent), intensity of exercise, and volume of exercise with BFR.

BFR along with low-load resistance training, cardio endurance training, and other activities that are generally recommended to improve muscular mass/strength are also associated with these adaptations in muscles.

The combination of Low-load Resistance Exercise with Body-Focused Rehabilitation (BFR) promotes greater strength adaptations and hypertrophy than the combination of Low-Load Resistance Exercise with BFR alone. Exercises that combine low load resistance with BFR can promote comparable levels of hypertrophy to those that combine high load resistance.

The review done by Vinolo-Gil and colleagues revealed that treatment with blood flow restriction appears to be helpful for neurological conditions without having side effects. Improvements have been shown in gait, quality of life, endurance, muscle strength, and limb functions.

Many studies done on the effect of BFRT on the lower limb in stroke patients, for an example the randomized trial done to compare low-intensity resistance training with BFR (LIRT-BFR) and high-intensity resistance training in stroke patients, results revealed that BFRT produced a significant improvement in lower limb strength, balance, gait, and depression No previous studies done on the effect of BFRT on upper limbs in post-stroke patients so This study aims to study the effect of Blood Flow Restriction training on motor function, strength, and Activity of daily living in stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* 30 ≥ years of age.
* The diagnosis of stroke
* Confirmed by cranial CT and/or MRI
* Hemipaises (weakness of one side of the body ), clear consciousness, stable vital signs

Exclusion Criteria:

* Uncontrolled hypertension
* Coronary artery disease
* Deep vein thrombosis
* Severe osteoarthritis
* Cognitive impairment, inability to cooperate
* Any severe musculoskeletal problem that prevented the participants from doing resistance training
* unstable complications related to heart, lung, and kidney diseases.
* Serious cognitive or audio-visual impairment
* Mini-Mental Scale Examination score, <24)

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-05-30 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Muscle power | at base line and after 8 weeks of tretment
  muscle power will be assessed using by Manual muscle test for shoulder and elbow flexor and extensor
2- Hand grip strength | at base line and after 8 weeks of tretment
  handgrip strength will be measured using (hand dynamometer ) Based on previous studies, the JAMAR® Hydraulic Hand Dynamometer has been widely used, and has been validated and reliable.
  1. The subject should sit with the back, pelvis, and knees as close to 90 degrees as possible.
  2. The shoulder is adducted and neutrally rotated, elbow at 90 degrees flexion, forearm neutral, wrist held between 0-15 degrees of ulnar deviation.
  3. A dynamometer is placed vertically on the forearm without support from the examiner or armrest.
  4. Three trials are taken to determine the maximum grip.
The Stroke Upper-Limb Capacity Scale | at base line and after 8 weeks of tretment
  The Stroke Upper-Limb Capacity Scale (SULCS) is a validated tool for upper extremity (UE) functional tasks, SULCS measures upper limb capacity, including basic arm capacities. There are ten items in the SULCS that represent meaningful tasks that relate to daily activities at home. The selection of these tasks was based on extensive interviews with rehabilitation physicians, occupational therapists, and physical therapists
Activity of daily living by Barthel Index | at base line and after 8 weeks of tretment
  Activity of daily living by Barthel Index Functional independence was assessed using the Barthel Index, validated for cerebrovascular diseases and elderly , The index analyzes 10 aspects: bowels, bladder, grooming, toilet use, feeding, transfer, mobility, dressing, stairs, and bathing. The total score ranges from 0 to 100 points. The higher the score, the greater the functional independence

SECONDARY OUTCOMES:
Modified Disability Arm Shoulder Hand | at base line and after 8 weeks of tretment
  Modified Disability Arm Shoulder Hand (QuickDASH), is a validated and widely used 11-item questionnaire that measures upper-extremity specific symptoms and disability
Patient satisfaction (PSQ 18) | at base line and after 8 weeks of tretment
  Patient Satisfaction Questionnaire Short Form PSQ18 was validated for use among various settings to measure Patient Satisfaction regarding medical services, it was shortened from substantially larger questionnaires while maintaining internal consistency and reliability ,there are seven dimensions of patient satisfaction with their doctors including (interpersonal manner, communication, financial aspect, time spent with the doctor), The response options required the patients to rate each item using a 5-point rating scale. A scale of 1-5 is used to rank the answers, with 1 equaling totally disagreeing and 5 equaling totally agreeing. A higher score indicates a better relationship between the patient and the doctor or a higher level of patient satisfaction

IPD SHARING:
Plan to Share IPD: No
the data could be used in future study